CLINICAL TRIAL: NCT01625078
Title: Observational Study of Baska Mask, a New Supraglottic Airway Device in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Laffey (Other)
Responsible Party: Sponsor-Investigator, John Laffey, Professor of Anaesthesia and Critical Care, University College Hospital Galway
Organization: University College Hospital Galway (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C.A.657
Record Dates: First submitted 2012-03-23; First posted 2012-06-21 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Baska Mask Efficacy and Safety in Children
Keywords: Baska Mask; Supraglottic airway device; Children; Pediatric
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Baska mask (Experimental)
  Interventions: Device: Placement and use of Baska mask

INTERVENTIONS:
Device: Placement and use of Baska mask — Use of Baska mask as a supraglottic airway during general anesthesia

SUMMARY:
The investigators wish to accumulate initial data on the performance and safety of the Baska mask in paediatric patient population.

ELIGIBILITY:
Inclusion Criteria:

* consent
* BMI 15-35
* weight over 30kg or age 8-16 yrs
* non-urgent surgery of planned duration up to 2 hrs

Exclusion Criteria:

* neck pathology
* previous or anticipated problems with the upper GI or upper airway
* increased risk of gastric aspiration
* expected difficult airway

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Device insertion success rate | within 30 minutes of induction of general anesthesia
device airway leak pressure | within 10 minutes of successful device placement
  the airway l;eak pressure is defined as the plateau airway pressure measured while the patient is apnoeic with the APL valve of the anaesthetic machine set to 35 cm H2O and the fresh gas flow set to 6 L/min

SECONDARY OUTCOMES:
airway stability | within 30 minutes of device placement
  the tidal volumes will be measured in different head positions and the leak fractions calculated.
ease of device placement | within 30 minutes of induction of general anesthesia
  the ease of device placement will be evaluated by Visual Analogue Scale
complications during the anesthetic | from the start of device insertion untill discharge from recovery, an expected average of 2 hours
  complications that may be related to the device use will be monitored including but not limited to desaturation episodes, laryngospasm, loss of airway, need to switch ot alternative device, blood staining on mask removal sore throat, dysphonia, dysphagia

CONTACTS AND LOCATIONS:
Overall Officials: Michael Scully, FFARCSI, Principal Investigator — UCHG
Locations (1):
- Galway University Hospitals, Galway, Galway, Ireland